CLINICAL TRIAL: NCT00729326
Title: Comparison of the Effect of Exenatide vs. Sitagliptin on 24-hour Average Glucose in Patients With Type 2 Diabetes on Metformin or a Thiazolidinedione
Brief Title: Comparison of the Effect of Exenatide Versus Sitagliptin on 24-hour Average Glucose in Patients With Type 2 Diabetes on Metformin or a Thiazolidinedione
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-US-GWCV
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; sitagliptin; Amylin; Lilly; metformin; thiazolidinedione
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: exenatide; Drug: sitagliptin; Drug: placebo
- Sequence B (Experimental)
  Interventions: Drug: exenatide; Drug: sitagliptin; Drug: placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection (5mcg or 10mcg), twice a day
  Other Names: Byetta
Drug: sitagliptin — oral administration (100mg), once a day in the morning
  Other Names: Januvia
Drug: placebo — subcutaneous injection (5mcg or 10mcg), twice a day
Drug: placebo — oral administration (100mg), once a day in the morning

SUMMARY:
This study is designed to compare the short-term effects and mechanisms of action of exenatide with those of sitagliptin when either is added to an oral agent(metformin or a thiazolidinedione [TZD]) in adult patients with type 2 diabetes mellitus(T2DM) with inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Has HbA1c 7.0% to 11.0%, at or within 4 weeks prior to Visit 1.
* Have a fasting glucose concentration <280 mg/dL at Visit 1
* Have been treated with a stable dose of immediate or extended release metformin for at least 60 days prior to screening OR TZD (rosiglitazone or pioglitazone) for at least 120 days prior to screening.
* Are between 18 and 70 years of age, inclusive.
* Have body mass index ≥25 kg/m2 and ≤45 kg/m2.
* Have a history of stable body weight (not varying by >10% for at least 3 months prior to screening).
* Can swallow oral study drug capsule, without splitting or crushing.

Exclusion Criteria:

* Female patients of childbearing potential (not surgically sterilized and between menarche and 1 year postmenopause) who meet any of the following criteria:

  * Are breastfeeding.
  * Test positive for pregnancy at the time of screening.
  * Intend to become pregnant during the study.
  * Have not practiced a reliable method of birth control (for example, use of oral contraceptives or Norplant®; diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices; partner with vasectomy; or abstinence) for 3 months prior to screening.
* Treated with any of the following medications:

  * Insulin, exenatide, pramlintide, sulfonylureas or meglitinides within 3 months of screening
  * Alpha-glucosidase inhibitor within 2 months of screening.
  * Drugs that directly affect gastrointestinal motility, including, but not limited to metoclopramide, cisapride, and chronic macrolide antibiotics.
  * Use of a drug for weight loss (for example, prescription drugs such as orlistat, sibutramine, phentermine, or similar over-the-counter medications) within 3 months prior to Visit 1.
  * Systemic corticosteroids by oral, intravenous, or intramuscular route within 2 months of screening.
* Have a history of renal transplantation or are currently receiving renal dialysis.
* Have obvious clinical signs or symptoms of liver disease or acute or chronic hepatitis.
* Have known active proliferative retinopathy or macular edema expected to need treatment with focal photocoagulation within 3 months.
* Have an active or untreated malignancy, or have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have had organ transplantation.
* Have received GLP-1 analogs other than exenatide or DPP-4 inhibitors within the previous 3 months.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (1):
- Research Site, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Followed By Sitagliptin: Exenatide 5mcg plus sitagliptin placebo for 1 week, then exenatide 10mcg plus sitagliptin placebo for 3 weeks. Followed by exenatide placebo plus sitagliptin 100mg for 1 week, then exenatide placebo plus sitagliptin 100mg for 3 weeks.
- Sitagliptin Followed By Exenatide: Exenatide placebo plus sitagliptin 100mg for 1 week, then exenatide placebo plus sitagliptin 100mg for 3 weeks. Followed by exenatide 5mcg plus sitagliptin placebo for 1 week, then exenatide 10mcg plus sitagliptin placebo for 3 weeks.
Period: Overall Study
Arm/Group | Exenatide Followed By Sitagliptin | Sitagliptin Followed By Exenatide
Started | 41 | 42
Completed | 31 | 33
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Subject Decision | 4 | 4
Not completed — Sponsor Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Followed By Sitagliptin | Sitagliptin Followed By Exenatide | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 37 | 71
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.10) | 53.5 (9.49) | 54.1 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 29 | 48
  Male | 22 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Time-averaged Glucose During a 24 Hour Period
Description: Change in time-averaged glucose during a 24-hour period from baseline to endpoint (i.e., time-averaged glucose over 24 hours at endpoint minus time-averaged glucose over 24 hours at baseline).
Time Frame: baseline and 8 Weeks
Population: The number of patients was determined based on 90% powering of the study. Analyses were based on data from all randomized patients receiving at least one dose of the study drug and completing at least one treatment period. For each patient, the missing data for some time points were imputed by linear interpolation.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Exenatide: Exenatide 5mcg plus sitagliptin placebo for 1 week, then exenatide 10mcg plus sitagliptin placebo for 3 weeks.
- Sitagliptin: Exenatide placebo plus sitagliptin 100mg for 1 week, then exenatide placebo plus sitagliptin 100mg for 3 weeks.
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 67 | 66
mg/dL | -41.65 (2.55) | -29.56 (2.58)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Null hypothesis: The 24-hour average glucose for exenatide was greater than or equal to that for sitagliptin after 4 weeks of treatment. The primary objective was to compare exenatide with sitagliptin on the time-averaged glucose during the 24-hour inpatient periods after 4 weeks of treatment; Test type: Superiority or Other; p < .001, ANCOVA — The p-values were not adjusted. The primary measure was change in 24-hour glucose without multiplicity adjustments for other analyses; Analyses for continuous variables adjusted for treatment, period, sequence, baseline of the continuous variable.Analysis method was Grizzle's model

2. Secondary Outcome: Change in Two-hour Postprandial Glucose After the Morning Meal
Description: Change in 2 hour post-prandial glucose after the morning meal from baseline to endpoint (i.e., glucose level 2 hours after the morning meal at baseline minus glucose level 2 hours after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in FAS who have both baseline and endpoint measurement; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
mg/dL | -108.35 (4.36) | -44.43 (4.40)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

3. Secondary Outcome: Change in Fasting Blood Glucose After the Morning Meal
Description: Change in fasting blood glucose after the morning meal from baseline to endpoint (i.e., fasting blood glucose after the morning meal at baseline minus fasting blood glucose after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in FAS who have both baseline and endpoint measurement; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 68 | 67
mg/dL | -28.93 (2.70) | -28.22 (2.71)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p = .766, ANCOVA

4. Secondary Outcome: Change in Postprandial Glucagon Area Under the Concentration-time Curve (AUC) After the Morning Meal
Description: Change in Postprandial Glucagon AUC after the morning meal (t=0 to 4 hours) (i.e., Glucagon AUC over the first 4 hours following the morning meal at baseline minus glucagon AUC over the first 4 hours following the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: pmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 68 | 67
pmol*hours/L | -29.60 (2.91) | -16.91 (2.93)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

5. Secondary Outcome: Change in Postprandial Glucagon AUC Excursion After the Morning Meal
Description: Change in postprandial glucagon AUC excursion after the morning meal (t=0 to 4 hours) (i.e., glucagon AUC excursion for 4 hours following the morning meal at baseline minus glucagon AUC excursion for 4 hours following the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: pmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 68 | 67
pmol*hours/L | -30.94 (2.12) | -14.93 (2.13)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

6. Secondary Outcome: Change in Postprandial Triglyceride AUC After the Morning Meal
Description: Change in postprandial triglyceride AUC after the morning meal (t=0 to 4 hours) (i.e., postprandial triglyceride AUC after the morning meal at baseline minus postprandial triglyceride AUC after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mg*hours/dL
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
mg*hours/dL | 0.83 (0.03) | 0.87 (0.03)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p = .117, ANCOVA

7. Secondary Outcome: Change in Postprandial Triglyceride AUC Excursion After the Morning Meal
Description: Change in postprandial triglyceride AUC excursion after the morning meal (t=0 to 4 hours) (i.e., postprandial triglyceride AUC excursion after the morning meal at baseline minus postprandial triglyceride AUC excursion after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mg*hours/dL
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
mg*hours/dL | -108.16 (8.38) | -41.39 (8.45)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

8. Secondary Outcome: Change in Postprandial C-peptide AUC After the Morning Meal
Description: Change in postprandial C-peptide AUC after the morning meal (t=0 to 4 hours) (i.e., postprandial C-peptide AUC after the morning meal at baseline minus postprandial C-peptide AUC after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: nmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
nmol*hours/L | -1.78 (0.28) | 0.25 (0.28)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

9. Secondary Outcome: Change in Postprandial C-peptide AUC Excursion After the Morning Meal
Description: Change in Postprandial C-peptide AUC excursion after the morning meal (t=0 to 4 hours) (i.e., postprandial C-peptide AUC excursion after the morning meal at baseline minus postprandial C-peptide AUC excursion after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: nmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
nmol*hours/L | -2.83 (0.29) | 0.14 (0.29)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

10. Secondary Outcome: Change in Postprandial Insulin AUC After the Morning Meal
Description: Change in postprandial insulin AUC after the morning meal (t=0 to 4 hours) (i.e., postprandial insulin AUC after the morning meal at baseline minus postprandial insulin AUC after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: pmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
pmol*hours/L | -396.12 (56.79) | -8.79 (57.32)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

11. Secondary Outcome: Change in Postprandial Insulin AUC Excursion After the Morning Meal
Description: Change in Postprandial insulin AUC excursion after the morning meal (t=0 to 4 hours) (i.e., postprandial insulin AUC excursion after the morning meal at baseline minus postprandial insulin AUC excursion after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: pmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
pmol*hours/L | -525.01 (58.77) | -34.83 (59.40)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

12. Secondary Outcome: Change in Postprandial Active GLP-1 AUC After the Morning Meal
Description: Change in Postprandial active GLP-1 AUC after the morning meal (t=0 to 4 hours) (i.e., postprandial active GLP-1 AUC after the morning meal at baseline minus postprandial active GLP-1 AUC after the morning meal at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: pmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
pmol*hours/L | -14.28 (3.12) | 47.37 (3.15)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

13. Secondary Outcome: Change in Postprandial Active GLP-1 AUC Excursion After the Monrning Meal
Description: Change in Postprandial active GLP-1 AUC excursion after the morning meal (t=0 to 4 hours) (i.e., postprandial active GLP-1 AUC excursion after the morning meal at baseline minus postprandial active GLP-1 AUC excursion after the morning meals at endpoint)
Time Frame: baseline and 8 Weeks
Population: All patients in the FAS who have both baseline and endpoint measurements; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: pmol*hours/L
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 69 | 68
pmol*hours/L | -14.04 (3.28) | 23.53 (3.31)
Statistical Analysis 1: Comparison: Exenatide vs Sitagliptin; Test type: Superiority or Other; p < .001, ANCOVA

14. Secondary Outcome: Percentage of Patients Experiencing Hypoglycemia (Baseline to Week 4)
Description: Percentage of patients experiencing minor hypoglycemia with a confirmed glucose <54mg/dL
Time Frame: 4 Weeks
Population: All patients in FAS
Measure: Number; unit: Percentage of patients
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 35 | 37
Percentage of patients | 2.9 | 2.7

15. Secondary Outcome: Episodes of Hypoglycemia (Baseline to Week 4)
Description: Number of episodes of hypoglycemia experienced during the first 4 weeks of the study
Time Frame: 4 weeks
Population: Full analysis set
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 35 | 37
episodes of hypoglycemia | 1 | 1

16. Secondary Outcome: Percentage of Patients Experiencing Hypoglycemia (Week 4 to Week 8)
Description: Percentage of patients experiencing minor hypoglycemia with a confirmed glucose <54mg/dL
Time Frame: 8 weeks
Population: All patients in FAS
Measure: Number; unit: Percentage of patients
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 35 | 34
Percentage of patients | 5.7 | 0.0

17. Secondary Outcome: Episodes of Hypoglycemia (Week 4 to Week 8)
Description: Number of episodes of hypoglycemia experienced between week 4 and week 8 of the study
Time Frame: 8 weeks
Population: All patients in FAS
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 35 | 34
episodes of hypoglycemia | 2 | 0

18. Secondary Outcome: Percentage of Patients Experiencing Hypoglycemia (Overall)
Description: Percentage of patients experiencing minor hypoglycemia with a confirmed glucose <54mg/dL
Time Frame: 4 weeks and 8 weeks
Population: All patients in FAS
Measure: Number; unit: Percentage of patients
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 70 | 71
Percentage of patients | 4.3 | 1.4

19. Secondary Outcome: Episodes of Hypoglycemia (Overall)
Description: Number of episodes of hypoglycemia experienced overall during the study
Time Frame: 4 weeks and 8 weeks
Population: All patients in FAS
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Exenatide | Sitagliptin
Number analyzed (Participants) | 70 | 71
episodes of hypoglycemia | 3 | 1

ADVERSE EVENTS:
Arm/Group | Exenatide | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/73
Other Adverse Events (participants affected / at risk) | 43/73 | 37/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=73) | Sitagliptin (N=73)
Anaphylactic reaction (Immune system disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=73) | Sitagliptin (N=73)
Nausea (Gastrointestinal disorders) | 27 | 12
Vomiting (Gastrointestinal disorders) | 15 | 4
Headache (Nervous system disorders) | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 7 | 8
Dizziness (Nervous system disorders) | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Abdominal discomfort (Gastrointestinal disorders) | 4 | 3
Asthenia (General disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days